CLINICAL TRIAL: NCT00930384
Title: A Case Control Study to Evaluate the Prevalence of Non-Alcoholic Fatty Liver Disease (NAFLD) Among Patients With Psoriasis
Brief Title: A Case Control Study Evaluating the Prevalence of Non-Alcoholic Fatty Liver Disease Among Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 030940
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-02

CONDITIONS: Psoriasis; Nonalcoholic Fatty Liver Disease
Keywords: psoriasis; fatty liver; metabolic syndrome
MeSH Terms: conditions — Psoriasis; Non-alcoholic Fatty Liver Disease; Fatty Liver; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Psoriasis group: All adult patients fulfilling inclusion criteria will be considered as cases in which psoriasis is detected and diagnosed by our principal investigator based on the clinical criteria accepted by American Academy of Dermatology. They will have an abdominal ultrasound performed by a radiologist to assess for the presence of nonalcoholic fatty liver disease. They will be referred to the research clinic to have a blood drawn.
- Control group: For every case an age, sex and body mass index (BMI range - kg/m2) matched control will be selected from the same dermatologic/radiologic clinic. The controls will be invited to voluntarily participate and informed consent will be obtained for performing ultrasonography and analytical tests to ensure the absence of manifest hepatic disease.

SUMMARY:
Main objectives

1. Establish the association of psoriasis and the presence of NAFLD in the patients with psoriasis attending dermatologic clinic center.

Secondary objective

1. Evaluate for the presence of other components metabolic syndrome in this group of patients including hypercholesterolemia, hypertension, obesity, and insulin resistance
2. Determine if there is an association between the extent and severity of psoriasis and the presence of NAFLD.
3. Identify an association between BMI and presence of NAFLD in people with psoriasis and use it as a predictive index for primary screening of NAFLD in psoriatic patients.

DETAILED DESCRIPTION:
Psoriasis is a common inflammatory disorder of the skin and in some patients the joints. Several reports have demonstrated a possible association between psoriasis and diabetes mellitus, obesity, hypertension, myocardial infarction, and heart failure.

Metabolic syndrome (MS) is a cluster of diabetes mellitus, hypertension, visceral obesity and hyperlipidemia and is thought to be caused by insulin resistance and the presence of a systemic inflammation which is evident by the increased level of inflammatory cytokines like TNF in this group of patients.

Non Alcoholic Fatty Liver Disease ( NAFLD) is the accumulation of fat vacuoles in the cytoplasm of hepatocytes and is believed to be the most common cause of chronic liver disease in developed countries. Currently, the metabolic syndrome has been found to be a strong predictor of NAFLD, and NAFLD is widely accepted to be the hepatic manifestation of the MS.

Since people with psoriasis have significantly higher rates of metabolic syndrome and regarding the fact that NAFLD is considered as the hepatic manifestation of MS, the purpose of this study is to determine the prevalence of NAFLD in subjects with psoriasis compared to the non -psoriatic population.

We have designed a case control study of patients who attend the dermatologic clinic at GWU with a clinical diagnosis of psoriasis. By performing a limited RUQ abdominal ultrasonography at the GWU hospital, we will be able to screen the patients with a possible diagnosis of NAFLD. Since NAFLD is a diagnosis of exclusion, those patients who have been screened positive for NAFLD, will be further evaluated for ruling out the other etiologies of fatty liver such as alcohol abuse and hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes from dermatologic or radiologic clinics, between the age 18 and 80 years who wish to voluntarily participate in the study and who have signed a written informed consent form to participate.

Exclusion Criteria:

* Alcohol intake > 30 g/day in males and > 20 g/day in females.
* Presence of chronic liver disease.
* Presence of the hepatitis B virus surface antigen or the presence of virus hepatitis C antibodies.
* History of methotrexate, systemic corticosteroid, amiodarone, tamoxifen, estrogens, and/or nifedipine.
* Pregnancy
* Subjects with conditions or diseases hindering data collection and follow up of the study such as incapacitating diseases, cognitive deterioration, institutionalized patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the Dermatology Clinic at George Washington University Hospital, Medical Faculty Associates.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of NAFLD in psoriasis patients as compared to controls, via hepatic ultrasonography. | After obtaining consent

SECONDARY OUTCOMES:
Evaluate for the presence of other components of the metabolic syndrome in the case and control group by measuring fasting blood glucose, blood pressure, waist circumference, and a lipid profile. | After consent is obtained
Identify a possible association between extent and severity of psoriasis, and the presence of NAFLD. | After consent is obtained

CONTACTS AND LOCATIONS:
Overall Officials: Alison Ehrlich, MD, MHS, Principal Investigator — GWU; Nadia Khati, MD, Study Chair — GWU; Monica Rengifo-Pardo, Study Chair — George Washington University
Locations (1):
- George Washington University Department of Dermatology, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Awosika O, Eleryan MG, Rengifo-Pardo M, Doherty L, Martin LW, Ehrlich A. A Case-control Study to Evaluate the Prevalence of Nonalcoholic Fatty Liver Disease Among Patients with Moderate-to-severe Psoriasis. J Clin Aesthet Dermatol. 2018 Jun;11(6):33-37. Epub 2018 Jun 1. PMID 29942422